CLINICAL TRIAL: NCT03371069
Title: Use of Methylphenidate in Children and Adolescents in France
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: 15FKU-MPH
Record Dates: First submitted 2016-09-07; First posted 2017-12-13 (Actual); Last update posted 2017-12-13 (Actual); Status verified 2017-11

CONDITIONS: Use of Methylphenidate in Children and Adolescents
Keywords: methylphenidate; drug utilisation study; pediatrics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- users of methylphenidate: Children and adolescents who are users of methylphenidate, 2010 to 2015
  Interventions: Other: users of methylphenidate

INTERVENTIONS:
Other: users of methylphenidate — Children and adolescents who are users of methylphenidate, 2010 to 2015

SUMMARY:
The use of methylphenidate in children and adolescents in France from 2010 to 2015

DETAILED DESCRIPTION:
To describe the use of methylphenidate in children and adolescents in France from 2010 to 2015

ELIGIBILITY:
Inclusion Criteria:

* children and adolescents (0-17 years)
* registered in the French Health Insurance Database from 2012-2015

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children and adolesents who are users of methylphenidate
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
use of methylphenidate over time | 6 years
  Describe of the use of methylphenidate over time to determine the impact of regulatory information of appropriate prescription conditions of use in September 2012

SECONDARY OUTCOMES:
Describe methylphenidate patterns of use over time | 6 years
  Pharmaceutical specialties (immediate or extended release forms) prescribed by type of delivery: initial or renewals.
  Profile of prescribers: hospital or private practice (general practitioners, specialists) depending on type of prescription (initial or renewal); geographical distribution of the prescribers Profile of patients: sex, average age and age classes (0-23 months, 2-5 years, 6-11 years, 12-17 years), socioeconomic status, long-lasting diseases status for psychosis, severe personality disorder, mental retardation.
  Pattern of methylphenidate use: duration of treatment, prolonged use, interruption of treatment.
Co-prescription of methylphenidate and non-psychostimulant psychotropic drugs | 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Florentia Kaguelidou, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hôpital Robert Debré, APHP, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided